CLINICAL TRIAL: NCT00548496
Title: A Proof-of-Concept Study Of SB-751689 In Men And Post-menopausal Women With A Fractured Distal Radius
Brief Title: A Phase IIa Study Of Men And Post-Menopausal Women With A Fractured Distal Radius
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR9108914
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Fracture Healing
Keywords: fractured wrist; Distal radial fracture,
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo-Controlled based on the two Intervention Groups below (Experimental): Placebo-Controlled based on the two Intervention Groups below.
  Interventions: Drug: SB-751689; Other: Placebo

INTERVENTIONS:
Drug: SB-751689 — SB-751689
Other: Placebo — Placebo to match

SUMMARY:
This is a study designed to test the safety and effectiveness of SB-751689 in the treatment of a distal radius fracture in post-menopausal women and men in comparison to placebo to determine if healing time of the fracture can be decreased.

ELIGIBILITY:
Inclusion Criteria:

fracture/broken distal radius bone conservative treatment including closed reduction and immobilization device men (>35 years <80) post-menopausal women (<80 yr)

Full In/Ex crit. and EPs as per Amendment 1, dated 7 Feb 08 Subject is willing and able to provide written informed consent Unilateral, extra-articular distal radius fractures AO/ASIF types 23-A2 and 23-A3 are permissible. (Arbeitsgemeinschaft für Osteosynthesefragen [AO]/ Association for the Study of Internal Fixation [ASIF]). Multiple fractures of bones, other than the limb with the distal radius fracture, are permissible if the subject can perform the protocol-required procedures.

Received conservative treatment of the distal radius fracture, including closed reduction and immobilization device (such as cast, splint, or brace) Ambulatory male and female subjects aged ≥35 to <80 years of age who have sustained a closed, unilateral, fracture of the distal radius no more than 5 days prior to randomization.

Females of non child-bearing potential defined as: >1 year postmenopausal, which can be >1 year of spontaneous amenorrhea or >1 year post surgical bilateral oophorectomy. Use follicle stimulating hormone [FSH] levels >40mIU/mL to confirm surgical postmenopausal status, where bilateral oophorectomy status is uncertain. Females of child-bearing potential must have a negative urine bhCG pregnancy test at the Screening visit and agree to practice acceptable highly effective methods of birth control throughout the duration of the study. Highly effective birth control methods include those preventative measures taken to avoid pregnancy that have a failure rate of less than 1% per year.

Subject who, in the opinion of the investigator, is willing and able to comply with the requirements of the protocol, including ability to understand patient reported outcomes (PRO) questionnaires

Exclusion Criteria:

-fracture occurred within 5 days of injury all AO B- and C-type prior fracture of the same wrist placement of hardware (pins and plates) diseases affecting bone metabolism inflammatory joint disease an increased risk of osteosarcoma malignant disease diagnosed within the previous 5 years (except resected basal cell cancer) past or current history of liver disease or known hepatic or biliary abnormalities treatment with fluoride (dose greater than 10 mg/day) within the previous 5 years for osteoporosis limitations of prior treatment with an oral bisphosphonate

Any treatment of a fractured distal radius that occurred more than 5 days after the fracture sustaining injury All B- and C-type fractures (intra-articular) according to AO Fracture classification or any distal radius fracture that would likely require open reduction and internal fixation. All additional fractures in the limb (including hand and humerus) with the distal radial fracture are excluded. Any fracture of the contralateral upper or lower arm, wrist or hand that would interfere with obtaining measurements on the dynamometer are excluded. Pathological (tumor-related) fractures Prior fracture of the same wrist as an adult Hardware including pins or plates in the wrist (either prior or current injury) History of or concurrent synovial pseudoarthrosis, congenital pseudoarthrosis, or active osteomyelitis History or concurrent diseases affecting bone metabolism (e.g., osteomalacia, hyperparathyroidism, etc.) History of skeletal immaturity Active disease or history of inflammatory joint disease (e.g., rheumatoid arthritis, lupus, psoriatic arthritis) that would interfere with imaging of the fracture Subjects receiving thyroid hormone replacement therapy should have thyroid stimulating hormone (TSH) levels measured.Subjects will be excluded if TSH levels are <0.1 or >10.0 mIU/L. However, subjects will not be excluded if TSH is in the range 0.1-4.5 mIU/L. If TSH is >4.5 to £10.0 mIU/L, measure T4 and exclude the subject only if the T4 is outside the normal range History of or active nephrolithiasis (kidney stones) Subjects at increased risk of osteosarcoma such as those with Paget's disease of bone or history of any prior external beam or implant radiation therapy involving the skeleton Malignant disease diagnosed within the previous 5 years (except resected basal cell cancer) Active or history of malabsorption (e.g., history of celiac disease, irritable bowel syndrome, or inflammatory bowel disease) Note: Subjects are not excluded because of previous or active gastrointestinal disease (i.e., prior history of non-recurrent peptic ulcer disease). Symptoms of dyspepsia, or Gastroesophageal Reflux Disease (GERD) must be able to be controlled by occasional use (not more than 3 doses per week) of a histamine-2 receptor antagonist Past or current history of liver disease or known hepatic or biliary abnormalities (with the exception of previously documented diagnosis of Gilbert's syndrome) Drug or alcohol abuse (past or current) within the previous 12 months A history of risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) A marked baseline prolongation of corrected QT interval (e.g., QTc interval ³450 msec on the Screening ECG corrected by either Bazett's or Fridericia's methodology) Surgical and medical conditions: Presence of the following conditions within 6 months prior to screening: myocardial infarction, coronary bypass surgery, coronary artery angioplasty, unstable angina, clinically evident congestive heart failure, cardiac pacemaker, or cerebrovascular accident: have currently known, suspected, or history of neurological diseases that affect the clinical assessments of healing; Cardiac arrhythmia: significant cardiac arrhythmias shown on screening ECG (as confirmed by eRT report), or a known or suspected history of significant cardiac arrhythmia's within 6 months prior to screening. i.e., pre-excitation syndromes, sinus pause >3 seconds, non-sustained ventricular tachycardia (³3 consecutive ectopic beats), sustained ventricular tachycardia (³30 consecutive ectopic beats), sustained supraventricular tachycardia (³30 consecutive ectopic beats), accessory pathway tachycardia, bradycardia (heart rate <50 beats per minute), atrial flutter, atrial fibrillation, ectopic pacemaker, sick sinus syndrome, atrioventricular block (second or third degree), or bundle branch block.

Any clinically relevant biological abnormality found and/or volunteered at screening (other than those related to the disease under investigation) which, in the opinion of the investigator, is clinically significant and would preclude safe participation in this study [e.g., human immunodeficiency virus infection and significant mental illness] Inability to swallow whole tablets Any previous treatment with strontium ranelate or intravenous bisphosphonate Any previous treatment with an oral bisphosphonate as follows: any treatment within the last 6 months; ≥ 1 month cumulative treatment within the last 12 months; ≥ 3 months cumulative treatment within the past 2 years, or ≥ 2 years cumulative treatment within the past 5 years Treatment with fluoride (dose greater than 10mg/day) within the previous 5 years for osteoporosis Treatment with PTH, PTH analogues or similar anabolic agent for osteoporosis within the last 2 years Treatment with other drugs affecting bone metabolism within the last 6 months prior to screening:Chronic systemic corticosteroid (e.g., glucocorticoid, mineralocorticoid) treatment of no more than 2 intra-articular injections within the past year or use of oral, parenteral, or long-term, high-dose inhaled corticosteroids. Treatment with any topical corticosteroid will not exclude the subject from participating; Hormones (e.g., estrogens/"natural estrogen preparations" [except for nonsystemic vaginal treatment], 19-norprogestins, selective estrogen receptor modulators [SERMs] such as raloxifene, anabolic steroids/androgens such as dehydroepiandrosterone [DHEA] or its sulfated form [DHEAS], nandrolone, tibolone, active vitamin D analogs/metabolites that are prescribed for the treatment of osteoporosis or other conditions such as 1,25-dihydroxy vitamin D [calcitriol] or 1-alpha-hydroxyvitamin D3 [1-alpha hydroxycholecalciferol], calcitonin); Calcineurin inhibitors (e.g., cyclosporine, tacrolimus) or methotrexate Contraindications to therapy with calcium or vitamin D Any subject who received treatment with the macrolide antibiotics: clarithromycin, erythromycin, telithromycin, and troleandomycin within 2 days prior to the Baseline visit Administration of any investigational drug within 90 days preceding the first dose of the study medication Current treatment with potent P-glycoprotein and/or potent CYP3A inhibitors is prohibited: Diltiazem and verapamil; any oral azole antifungal (e.g., ketoconazole, itraconazole, fluconazole); Cyclosporine or oral tacrolimus; Ritonavir; Quinidine; Nefazodone Concomitant therapy with proton pump inhibitors (e.g., esomeprazole, lansoprazole, omeprazole, pantoprazole, and rabeprazole) is prohibited. Daily, chronic use (>3 doses per week) of histamine-2 receptor antagonists (e.g., cimetidine, famotidine, nizatidine, and ranitidine) is prohibited. Antacids should not be administered within 2 hours (before or after) administration of study medication.

Vitamin A in excess of 10,000 IU per day, heparin, lithium, or anticonvulsant medications (except benzodiazepines) Current therapy with digoxin Subjects taking daily, long-term (i.e., > 1 year) non-steroidal anti-inflammatory drugs (NSAIDs) for diseases such as inflammatory arthritis are excluded. The use of low dose aspirin for prevention of heart disease is permitted. Short term use of NSAIDs is permitted for acute pain management but the use of alternative, non-NSAIDs is encouraged Total serum calcium levels outside the local laboratory reference range at the Screening visit Liver chemistries (aspartate aminotransferase [AST], alanine aminotransferase [ALT], or total bilirubin) exceeding 2-fold the upper limit of the local laboratory reference range at the Screening visit Glomerular filtration rate (GFR) <35 mL/min as calculated by the Modification of Diet in Renal Disease (MDRD) equation as follows: GFR (mL/min/1.73 m2) = 186 x (Serum creatinine mg/dL)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if African American) (conventional units) Women who are pregnant or breast-feeding are not allowed in the study. Females of child-bearing potential must have a negative urine bhCG pregnancy test at the Screening and Randomization visit and agree to practice acceptable highly effective methods of birth control through the duration of the study and for 4 weeks following the last dose of study medication. Highly effective birth control methods include those preventative measures taken to avoid pregnancy that have a failure rate of less than 1% per year.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-09-20 (Actual); Primary Completion 2008-11-26 (Actual); Study Completion 2008-11-26 (Actual)

PRIMARY OUTCOMES:
Data from the study will be used to determine if fracture healing time at 16 weeks is decreased in patients receiving SB-751689 and will determine future studies. | 16 Weeks

SECONDARY OUTCOMES:
Radiographic, functional, and quality of life assessments. | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- Argentina (8):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Naciones Unidas 346, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Juan
- Australia (3):
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Geelong, Victoria
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, Hong Kong, Hong Kong
- Netherlands (3):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leiden
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Africa (2):
  - GSK Investigational Site, Bryanston
  - GSK Investigational Site, Pinelands
- GSK Investigational Site, Seoul, South Korea
- Spain (3):
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Kungälv
  - GSK Investigational Site, Mölndal
- Taiwan (2):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Taichung
- United Kingdom (2):
  - GSK Investigational Site, Rhyl, Flintshire
  - GSK Investigational Site, Edinburgh, Midlothian

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Fitzpatrick LA, Smith PL, McBride TA, Fries MA, Hossain M, Dabrowski CE, Gordon DN. Ronacaleret, a calcium-sensing receptor antagonist, has no significant effect on radial fracture healing time: results of a randomized, double-blinded, placebo-controlled Phase II clinical trial. Bone. 2011 Oct;49(4):845-52. doi: 10.1016/j.bone.2011.06.017. Epub 2011 Jun 30. PMID 21742071
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: CR9108914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: CR9108914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CR9108914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: CR9108914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CR9108914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: CR9108914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: CR9108914 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register